CLINICAL TRIAL: NCT03953105
Title: Electronic Pediatric Emergency Ruler vs the Broselow Tape in a Simulated Pediatric Emergency Scenario
Brief Title: Electronic Pediatric Emergency Ruler vs the Broselow Tape.
Acronym: ePERvsBT
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ePER vs BT
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Time Until Identification of Defined Parameter
Keywords: Weight estimation; Patient safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Resusci Baby: Resusci Baby used for the simulated emergency scenario
  Interventions: Device: ePER; Device: BT
- Ambu® Junior: Ambu® Junior used for the simulated emergency scenario
  Interventions: Device: ePER; Device: BT

INTERVENTIONS:
Device: ePER — usind the ePER for weight estimation and suggestion of the defined parameter
Device: BT — usind the BT for weight estimation and suggestion of the defined parameter

SUMMARY:
Comparison of two different pediatric emergency rulers for length-based body weight estimation in pediatric emergencies.

Primary outcome is the time needed to identify four defined parameters from the pediatric emergency rulers during a low-fidelity pediatric emergency scenario (cardiac arrest). Secondary outcome is the correctness of the identified parameters and the percentage deviation from the correct value.

DETAILED DESCRIPTION:
Medical team members (Paramedics, EMT) of Schutz und Rettung Zurich, Zurich Switzerland were asked to participate in this study. If they were not familiar with one of the three devices written informed consent was obtained and the participant included in this study. This exclusion criteria was necessary to prevent a bias by already knowing where to find the information of interest.

The pediatric emergency rulers investigated were the electronic Pediatric Emergency Ruler (ePER) and the Broselow Tape (BT)

All participants were instructed for the use of the two pediatric emergency rulers and were given time to practice with each device using one training manikin (Sim-Baby)

After they felt comfortable using the devices the participants were randomly assigned to use each device only once with one of two different manikins:

Resusci Baby, Laerdal/Dräger Medical Switzerland AG, Liebefeld, Switzerland Ambu® Junior, Ambu® GmbH, Bad Nauheim, Germany

Each manikin was only used once for the same participant. This guaranteed that the participants were blinded for the manikins.

The low-fidelity pediatric emergency scenario simulated was a cardiac arrest and the participants were asked to identify the following information from the pediatric emergency rulers:

Estimated body weight Joule suggested for defibrillation Recommended epinephrine dose Suggested endotracheal tube size

Participants stood aside from the manikin with a pediatric emergency ruler in their hand. After they stated they were ready, the facilitator started a countdown from three and gave the command to start. This setting was identical for all two pediatric emergency rulers and all two manikins. The time until each parameter was identified and the value of the parameter were recorded.

Primary outcome was the time needed to identify the four above defined parameters. Secondary outcome was the correctness of the identified parameters and the percentage deviation from the correct value.

ELIGIBILITY:
Inclusion Criteria:

* Medical team members (Paramedics, EMT) of Schutz und Rettung Zurich, Zurich, Switzerland
* Written informed consent

Exclusion Criteria:

* Having worked with one of the pediatric emergency rulers and knowing where to find the defined parameters

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Medical team members (Paramedics, EMT) of Schutz und Rettung Zurich, Zurich, Switzerland
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Time to identification | During simulation, approximately 30 minutes
  Time needed to identify the four defined parameters

SECONDARY OUTCOMES:
Correctness | During simulation, approximately 30 minutes
  Correctness of the identified Parameter. The from the participant identified value is compared with the per value defined correctly based on the manikin size.
Percentage deviation | During simulation, approximately 30 minutes
  If the Parameter was identified incorrectly, a percentage deviation of the identified value from the correct value will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Schmidt, MD, Principal Investigator — Department of Anaesthesia and Children's Research Centre, University Children's Hospital, Zurich, Switzerland
Locations (1):
- University Childrens Hospital, Department of Anaesthesia and Children's Research Centre, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided